CLINICAL TRIAL: NCT06681220
Title: Biomarker Directed Trial of Temozolomide and Stenoparib in Relapsed SCLC
Acronym: Relapsed SCLC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPLP-002-24S; 14094144/CX002801-01A1 (Other Grant/Funding Number: VA Clinical Science Research & Development)
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Small Cell Lung Cancer; Recurrent Small Cell Lung Cancer
Keywords: Phase 2; Small Cell Lung Cancer; Biomarker
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — stenoparib; Temozolomide; PM 01183

STUDY DESIGN:
Intervention Model Description: The study will include 9 participants for the safety evaluation of the Stenoparib+TMZ group and 5 participants for the standard of care Lurbinectedin safety group. We will first determine safety dose for the experiment arm which, will include 3 groups with 3 participants in each group. Three doses of Stenoparib will be evaluated for toxicity. The initial starting dose of Stenoparib will be 200mg po QD. Once the maximum tolerated dose has been determined, participants will be assigned to one of the two groups in the phase 2 portion. Participants will receive either a combination of oral Stenoparib at the highest tolerated dose with oral Temozolomide 40mg daily or standard of care Lurbinectin for 21-day cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Study Drug Combination (Experimental): Biomarker positive patients will be randomized 2:1 to study drug (Stenoparib at the recommended phase 2 dose +TMZ 40mg/day daily) or (Standard of Care) Lurbinectedin 3.2mg/m2 one-hour intravenous (IV) infusion each cycle x21 days until disease progression or intolerable toxicity
  Interventions: Combination Product: Stenoparib/Temozolomide
- Standard of Care (Active Comparator): Lurbinectedin 3.2mg/m2 one-hour intravenous (IV) infusion each cycle x21 days until disease progression or intolerable toxicity
  Interventions: Drug: Lurbinectedin
- Biomarker Negative Standard of Care (Active Comparator): Lurbinectedin 3.2mg/m2 one-hour intravenous (IV) infusion each cycle x21 days until disease progression or intolerable toxicity
  Interventions: Drug: Lurbinectedin
- Safety lead-in (Experimental): Biomarker positive patients will be assigned to one of three doses of Stenoparib (200mg po qd, 200mg po BID, and 200mg in am and 400mg in pm). The initial starting dose will be the 200 mg po QD orally daily for 21 days.
  Interventions: Combination Product: Stenoparib/Temozolomide

INTERVENTIONS:
Combination Product: Stenoparib/Temozolomide — Stenoparib at the recommended phase 2 dose +Temozolomide 40mg/day daily will be given in combination x21 days each cycle
  Other Names: Stenoparib/TEMODAR
  Arms: Study Drug Combination
Drug: Lurbinectedin — Lurbinectedin 3.2mg/m2 one-hour intravenous (IV) infusion x 21 days each cycle
  Other Names: Zepzelca
  Arms: Biomarker Negative Standard of Care; Standard of Care
Combination Product: Stenoparib/Temozolomide — Patients will be assigned to one of three doses of Stenoparib (200mg po qd, 200mg po BID, and 200mg in am and 400mg in pm). The initial starting dose will be the 200 mg po QD orally daily for 21 days.
  Other Names: Stenoparib/TEMODAR
  Arms: Safety lead-in

SUMMARY:
Randomized phase 2, multicenter, biomarker directed clinical trial with a safety lead-in to assess the efficacy of Stenoparib plus Temozolomide (TMZ) in relapsed Small Cell Lung Cancer patients. Participants will receive either a combination of oral Stenoparib at the highest tolerated dose with oral Temozolomide 40mg daily or standard of care Lurbinectedin for 21-day cycles. The Dose limiting toxicity period will be 1 cycle of 21 days. This study will explore if the biomarkers the investigators test predict sensitivity to the combination of Stenoparib plus TMZ and therefore leads to a better treatment response. There are two potential tests of biomarkers that can predict who would benefit from the oral combination of Stenoparib with Temozolomide (TMZ), but they have not been evaluated. This study will test for this sensitivity using a biomarker (found in the blood that may be related to how a person reacts to a drug). The study will include 9 participants for the safety evaluation of the Stenoparib+TMZ group and 5 participants for the standard of care Lurbinectedin safety group. We will first determine safety dose for the experiment arm which, will include 3 groups with 3 participants in each group. Three doses of Stenoparib will be evaluated for toxicity. The initial starting dose of Stenoparib will be 200mg po QD. Once the maximum tolerated dose has been determined, participants will be assigned to one of the two groups in the phase 2 portion. Group 1 will be patients that test negative for the biomarker and will receive treatment with Lurbinectedin as per standard of care guidelines. Group 2 will be patients that test positive for the biomarker that will be randomly assigned to either the combination of Stenoparib plus Temozolomide (TMZ) or Lurbinectedin.

DETAILED DESCRIPTION:
Randomized phase 2, multicenter, biomarker directed clinical trial with a safety lead-in to assess the efficacy of Stenoparib plus Temozolomide (TMZ) in relapsed Small Cell Lung Cancer patients. Participants will receive either a combination of oral Stenoparib at the highest tolerated dose with oral Temozolomide 40mg daily or standard of care Lurbinectedin for 21-day cycles. The Dose limiting toxicity period will be 1 cycle of 21 days. This study will explore if the biomarkers the investigators test predict sensitivity to the combination of Stenoparib plus TMZ and therefore leads to a better treatment response. There are two potential tests of biomarkers that can predict who would benefit from the oral combination of Stenoparib with Temozolomide (TMZ), but they have not been evaluated. This study will test for this sensitivity using a biomarker (found in the blood that may be related to how a person reacts to a drug). The study will include 9 participants for the safety evaluation of the Stenoparib+TMZ group and 5 participants for the standard of care Lurbinectedin safety group. We will first determine safety dose for the experiment arm which, will include 3 groups with 3 participants in each group. Three doses of Stenoparib will be evaluated for toxicity. The initial starting dose of Stenoparib will be 200mg po QD. Once the maximum tolerated dose has been determined, participants will be assigned to one of the two groups in the phase 2 portion. Group 1 will be patients that test negative for the biomarker and will receive treatment with Lurbinectedin as per standard of care guidelines. Group 2 will be patients that test positive for the biomarker that will be randomly assigned to either the combination of Stenoparib plus Temozolomide (TMZ) or Lurbinectedin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of consent.
* Histological or cytological diagnosis of extensive-stage small cell lung cancer.
* Patients must have received one prior line of systemic therapy.

  * Patients must have received first-line therapy with Carboplatin and Etoposide.

    * If patient is re-treated with Carboplatin and Etoposide at least 6 months or more after first regimen, this will still be considered one line of
    * treatment and they will qualify for this trial.
  * Patients could have received immunotherapy in combination with the chemotherapy regimen.
  * Patients who have received Tarlatamab as second line treatment are allowed.
* ECOG Performance status 0-2.
* Measurable disease as per RECIST v1.1 (NOTE: Previously irradiated lesions are eligible as a target lesion only if there is documented progression of the lesion after irradiation).
* Adequate bone marrow, liver, and renal function, as assessed by the following laboratory requirements:

  * ANC 1.5
  * Platelets 100 × 109/L
  * Hemoglobin 9 g/dL or 5.6 mmol/L
  * Aspartate transaminase and alanine transaminase 2.5 × upper limit of normal (ULN), <5× in patients with known liver metastases
  * Serum total bilirubin 1.5 × ULN, 1.5-3.0 × ULN may be included appropriate starting dose adjustment to 200 mg daily.
  * Creatinine <1.5 × ULN or estimated glomerular filtration rate (GFR) 50 ml/min by Cockcroft-Gault. Depending on scenario, GFR 30-49 can be --permissible.
* Women of child-bearing potential must not be pregnant or breastfeeding and must have a negative pregnancy test within 72 hours of cycle 1 Day 1.
* Male and female subjects of child-bearing potential must agree to use a double-barrier method of birth control from the screening visit through 180 days after the last dose of study drug.
* Male subjects of child-bearing potential must agree to use a double-barrier method of birth control including use a male condom (and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak) and must agree to refrain from donating sperm from screening visit through at least 90 days after the last dose of study drug.
* Previously treated or asymptomatic brain metastases are allowed.

Exclusion Criteria:

* Unstable or clinically significant concurrent medical condition, psychiatric illness or social situation that would, in the opinion of the investigator, jeopardize the safety of a subject and/or their compliance with the protocol.
* Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy. (Suppressive therapy for chronic infections allowed, for example: Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed. Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy.)
* Prior exposure to lurbinectedin, TMZ or stenoparib.
* Pregnant or breastfeeding.
* Clinical significant cardiovascular disease (ie active)
* Subject with known hypersensitivity to Stenoparib components
* Subject with known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) are excluded.
* Subject with QTc interval 470 for females, or 450 for males per electrocardiogram (EKG) at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Through study completion up to 2 years.
  According to response evaluation criteria in solid tumors RECIST 1.1(imaging criteria or progression or patient death).
Recommended Phase 2 dose | Through end of cycle 1 (21 days)
  Defined as the recommended dose of Stenoparib for phase 2

SECONDARY OUTCOMES:
Disease control rate (DCR) | Through study completion up to 2 years.
  Defined as Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) per RECIST 1.1.
Overall Survival (OS) | Through study completion up to 2 years.
  Will be measured from Day 1 of treatment until death from any cause.
Overall response rate (ORR) | Through study completion up to 2 years.
  Defined as complete response (CR) + partial response (PR) per RECIST 1.1 criteria.
Treatment Toxicities | Through study completion up to 2 years.
  As defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Progression Free Survival (PFS) | Through study completion up to 2 years.
  Compare PFS between biomarker positive and biomarker negative patient receiving Lurbinectedin.

CONTACTS AND LOCATIONS:
Overall Officials: Shadia Jalal, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (11):
- United States (11):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Robley Rex VA Medical Center, Louisville, KY, Louisville, Kentucky
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No